CLINICAL TRIAL: NCT00294320
Title: Pilot Study to Evaluate Two Different Non-invasive Techniques to Monitor the Clearance of Actinic Keratosis Lesions (Clinical and Sub-clinical), When Treated With Aldara 5% (Imiquimod) Cream
Brief Title: Evaluation of Two Different Non-invasive Techniques to Monitor the Clearance of Actinic Keratosis Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Dr Elena Rizova MD. PhD Medical & Scientific Affairs Europe & MENA, Laboratoires 3M Santé
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1517-IMIQ
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2008-09

CONDITIONS: Actinic Keratosis
Keywords: Aldara; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 250mg of Imiquimod cream application once daily 3 times per week.
  Interventions: Drug: Aldara (Imiquimod)
- 2 (Placebo Comparator): 250mg vehicle cream for application once daily 3 times per week.
  Interventions: Other: Vehicle cream

INTERVENTIONS:
Drug: Aldara (Imiquimod) — 250mg of Imiquimod cream for application once daily 3 times per week.
  Arms: 1
Other: Vehicle cream — 250mg vehicle cream for application once daily 3 times per week.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the performance of two techniques to monitor the clearance of AK lesions when treated with Aldara 5% cream.

DETAILED DESCRIPTION:
Each technique will be assessed by comparison of lesion counts (clinical and sub-clinical) revealed by the techniques, at start and end of the study and those demonstrated during treatment. In addition a qualitative assessment of each technique will be made for performance and ease of use.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 clinically typical, visible, discrete, nonhyperkeratotic, nonhypertrophic AK lesions
* Free of any significant findings (e.g tattoos) in the potential application site area.
* Willing to discontinue sun-tanning and use of sunbed/sun parlour use
* Willing to stop use of moisturisers, body oils, and over the counter retinol products or products containing alpha or beta hydroxyacids in the treatment or surrounding area.
* Willing ot withhold sunscreen and/or moisturiser use for 24 hours prior to each clinical assessment

Exclusion Criteria:

* Evidence of unstable or uncontrolled clinically significant medical condition.
* Any dermatological disease and or condition in the treatment of the surrounding area that may be exacerbated by treatment with imiquimod.
* Currently participating in another clinical study or have completed another study within an investigational drug within the past 30 days.
* Have active chemical dependency or alcoholism
* Have know allergies to any excipient or study cream
* Have received previous treatment with imiquimod for any indication within the treatment area.
* Known to be affected by porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To compare the performance of two techniques to monitor the clearance of AK lesions (clinical and subclinical) when treated with Aldara 5% cream by comparison of lesion counts. | 8 weeks after the end of treatment

SECONDARY OUTCOMES:
To obtain histological confirmation of the diagnosis of the lesions demonstrated by biopsy. | 8 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Ortonne, Professor, Principal Investigator — CPCAD, Hopital L'Archet 2
Locations (1):
- Hopital L'Archet 2, Nice, Cedex 3, France